CLINICAL TRIAL: NCT07183982
Title: Effectiveness of a Multidisciplinary Rehabilitation Program for Treatment-Resistant Psychotic Patients in a Forensic Psychiatric Setting: A Comparative Study
Brief Title: Multidisciplinary Rehabilitation Program for Treatment-Resistant Psychotic Forensic Patients: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Sara Habib, Principal Investigator, Oman Ministry of Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MoH/CSR/24/28654
Record Dates: First submitted 2025-08-28; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Schizophenia Disorder; Forensic Psychiatric Patients
Keywords: Rehabilitation; Resistant Schizophrenia; Forensic
MeSH Terms: interventions — Rehabilitation; Art Therapy

STUDY DESIGN:
Intervention Model Description: This quasi-experimental, non-randomized parallel-group study evaluates a 6-month multidisciplinary rehabilitation program for forensic psychiatric inpatients with treatment-resistant psychotic symptoms at Al Masarra Hospital. Twenty patients will be allocated by convenience sampling to an intervention group (n=10) or control group (n=10). The intervention integrates psychodynamic group therapy, art therapy, music therapy, and cognitive stimulation (4-5 hrs/week), while controls receive standard physiotherapy and occupational therapy (3-4 hrs/week). PANSS and MoCA will be administered at baseline and post-intervention by blinded assessors. Data will be analyzed using Wilcoxon Signed-Rank and Mann-Whitney U tests, with effect sizes reported via Cliff's Delta. The null hypothesis is that there will be no significant differences in psychotic symptoms or cognition between groups post-intervention. outcomes may support rehabilitation importance in forensic settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Multidisciplinary Rehabilitation Arm (Experimental): 10 forensic psychiatric patients selected via convenience sampling from the forensic department of Al Masarra Hospital. All participants are diagnosed with treatment-resistant psychotic disorders and exhibit persistent cognitive, social, and functional deficits despite receiving pharmacological treatment. The patients included in this group match the inclusion criteria.
  This group is enrolled in a 6-month structured multidisciplinary rehabilitation program that integrates four distinct therapeutic modalities, each targeting a different domain of recovery: psychodynamic group therapy, art therapy, music therapy, and cognitive stimulation beside the tradition rehabilitation done (physiotherapy and occupational therapy. The integration of these therapies is designed to address the residual psychotic symptoms, cognitive, functional, emotional and relational impairments of the patients with resistant psychotic symptoms, which are often neglected in standard rehabilitation approaches.
  Interventions: Diagnostic Test: MoCA: Montreal Cognitive Assessment (MoCA) and Positive and Negative Syndrome Scale (PANSS); Behavioral: Rehabilitation program in the form of : psychodynamic group therapy, music and art therapy , cognitive stimulation techniques
- Control Group: Standard Rehabilitation Arm (Experimental): The control group consists of another 10 forensic psychiatric patients selected from the same department using the same inclusion criteria and sampling method. These patients are also diagnosed with treatment-resistant psychotic disorders and have longstanding impairments in cognition, functioning, and social interaction. However, instead of receiving the enhanced multidisciplinary program, they participate in the existing standard rehabilitation services provided at Al Masarra Hospital. This group serves as the comparison arm (control group) in this comparative experimental study.
  The standard rehabilitation program primarily includes physiotherapy and occupational therapy, both of which are routinely available within the hospital's forensic unit. These therapies aim to maintain physical health and promote basic functional independence in hospitalized patients with severe mental illness.
  Interventions: Diagnostic Test: MoCA: Montreal Cognitive Assessment (MoCA) and Positive and Negative Syndrome Scale (PANSS)

INTERVENTIONS:
Diagnostic Test: MoCA: Montreal Cognitive Assessment (MoCA) and Positive and Negative Syndrome Scale (PANSS) — MoCA: A 30-point screening tool assessing attention, memory, language, visuospatial and executive functions; quick and sensitive to mild cognitive deficits.
  PANSS: A 30-item scale rating positive, negative, and general psychopathology symptoms in psychotic disorders; widely used to track severity and change.
Behavioral: Rehabilitation program in the form of : psychodynamic group therapy, music and art therapy , cognitive stimulation techniques — Participants received a structured 6-month program designed to address persistent psychotic symptoms and associated deficits. The intervention included:
  Art Therapy: Weekly sessions promoting self-expression, emotional regulation, and enhancement of social interaction.
  Cognitive Stimulation: Structured group exercises aimed at improving attention, memory, executive functions, and problem-solving.
  The program was delivered by a multidisciplinary team in a group of 10 patients, ensuring active participation, individualized support, and integration of therapeutic modalities.
  Arms: Intervention Group: Multidisciplinary Rehabilitation Arm

SUMMARY:
This study employs a quasi-experimental design to evaluate the effectiveness of a 6-month multidisciplinary rehabilitation program integrating psychodynamic group therapy, art therapy, music therapy, and cognitive stimulation compared to standard rehabilitation (physiotherapy and occupational therapy). It will be done between a group of a total of 20 patients are divided into an intervention group and a control group from the forensic psychiatric department in Al Masarra Hospital.

DETAILED DESCRIPTION:
Forensic psychiatric patients with treatment-resistant psychotic symptoms often experience persistent cognitive, functional, and social deficits, posing significant challenges to rehabilitation. Traditional approaches may not adequately address these complex needs, highlighting the importance of innovative, multidisciplinary interventions. This study employs a quasi-experimental design to evaluate the effectiveness of a 6-month multidisciplinary rehabilitation program integrating psychodynamic group therapy, art therapy, music therapy, and cognitive stimulation compared to standard rehabilitation (physiotherapy and occupational therapy). A total of 20 patients are divided into an intervention group (n=10) and a control group (n=10) using convenience sampling from the forensic psychiatric department in Al Masarra Hospital. Data is collected using the Positive and Negative Syndrome Scale (PANSS) to assess psychotic symptoms and the Montreal Cognitive Assessment (MoCA) to evaluate cognitive function, administered at baseline and post-intervention. Data is analyzed using descriptive statistics (median, interquartile range) and non-parametric tests, including the Wilcoxon Signed-Rank Test for within-group comparisons and the Mann-Whitney U Test for between-group comparisons. Effect sizes are calculated using Cliff's Delta to assess the practical significance of the findings. The null hypothesis states that there will be no significant difference in PANSS and MoCA scores between the intervention and control groups post-intervention. If the null hypothesis is rejected, the findings will provide evidence for integrating creative and psychotherapeutic interventions into forensic psychiatric rehabilitation, offering a scalable model for similar settings.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic psychotic disorder (e.g., schizophrenia or schizoaffective disorder) confirmed by psychiatric assessment and medical records.
2. Presence of residual psychotic symptoms (positive symptoms such as hallucinations, delusions; and/or negative symptoms such as blunted affect, social withdrawal) despite ongoing psychotropic treatment.
3. Medically stable and deemed suitable for participation by the treating psychiatrist or healthcare team.
4. Patients who provide informed consent to participate in the rehabilitation program and research study.

Exclusion Criteria:

1. Acute medical or psychiatric conditions requiring immediate intervention.
2. Developmental or intellectual disabilities that significantly impair participation in the rehabilitation program or assessments.
3. Current substance dependence that would interfere with participation.
4. Significant risk of harm to self or others, based on clinical assessment or history of violence/aggression.
5. Contraindications to specific rehabilitation program components (e.g., physical exercise, group activities) as determined by medical evaluation.
6. Inability to comprehend study requirements or provide informed consent due to language barriers, cognitive impairment, or other factors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychotic Symptoms Measured by the Positive and Negative Syndrome Scale (PANSS) | Baseline (pre-intervention) and 6 months (post-intervention).
  Psychotic symptom severity will be assessed using the Positive and Negative Syndrome Scale (PANSS). Scores range from 30 to 210, with higher scores indicating greater severity. The unit of measure is score change from baseline to post-intervention.

SECONDARY OUTCOMES:
Change in Cognitive Function Measured by the Montreal Cognitive Assessment (MoCA) scale | Baseline (pre-intervention) and 6 months (post intervention).
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) scale. Scores range from 0 to 30, with higher scores indicating better cognitive performance. The unit of measure is score change from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sara A. Habib, Specialist, Principal Investigator — Al Massara Hospital,MOH Oman
Locations (1):
- Al Massara Hospital, Muscat, Muḩāfaz̧at Masqaţ, Oman